CLINICAL TRIAL: NCT00533923
Title: Nonmyeloablative Allogeneic Stem Cell Transplantation From HLA-Matched Unrelated Donor for the Treatment of Hematologic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, David McDermott, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002P000219
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: AML; ALL; CLL; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma; Hodgkin's Lymphoma; Multiple Myeloma; Aplastic Anemia; Myeloproliferative Disorder
Keywords: Nonmyeloablative Allogeneic Stem Cell Transplantation; mini-transplant; AML; ALL; CML; CLL; Myelodysplastic syndrome; Relapsed non-Hodgkin's or Hodgkin's lymphoma; Relapsed multiple myeloma; Aplastic anemia; Myeloproliferative disorder; GM-CSF; Cyclosporin; Fludarabine (FLUDARA); Cyclophosphamide; CAMPATH-1H; GVHD; CMV; AML in first remission, first relapse or subsequent remission; ALL in first relapse, second or subsequent remission; ALL in first remission, in a high-risk category; Aplastic anemia characterized by ANC< 1000 and/or platelets < 30 without transfusional support; Myeloproliferative disorder (P Vera, CMML, ET)
MeSH Terms: conditions — Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Anemia, Aplastic; Myeloproliferative Disorders; Neoplasm Metastasis | interventions — Cyclophosphamide; fludarabine; Cyclosporine; Alemtuzumab; Granulocyte-Macrophage Colony-Stimulating Factor; fludarabine phosphate; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cyclophosphamide; Fludarabine; Cyclosporin; CAMPATH-1H (Alemtuzumab); GM-CSF — intravenous
  Other Names: Cytoxan;; Fludara;; Leukine;

SUMMARY:
Allogeneic stem cell transplantation may provide long-term remissions for some patients with hematological malignancies. However, allogeneic transplantation is associated with a significant risk of potentially life threatening complications due to the effects of chemotherapy and radiation on the body and the risks of serious infection. In addition, patients may develop a condition called Graft versus host disease that arises from an inflammatory reaction of the donor cells against the recipient's normal tissues. The risk of graft versus host disease is somewhat increased in patients who are receiving a transplant from an unrelated donor.

One approach to reduce the toxicity of allogeneic transplantation is a strategy call nonmyeloablative or "mini" transplants. In this approach, patients receive a lower dose of chemotherapy in an effort to limit treatment related side effects. Patients undergoing this kind of transplant remain at risk for graft versus host disease particularly if they receive a transplant from an unrelated donor. The purpose of this research study is to examine the ability of a drug called CAMPATH-1H to reduce the risk of graft versus host disease and make transplantation safer. CAMPATH-1H binds to and eliminates cells in the system such as T cells that can cause graft versus host disease (GvHD). As a result, earlier studies have shown that patients who receive CAMPATH-1H with an allogeneic transplant have a lower risk of GvHD. In the present study, we will examine the impact of treatment with CAMPATH-1H as part of an allogeneic transplant on the development of GvHD and infection. In addition, we will study the effects of CAMPATH-1H on the immune system by testing blood samples in the laboratory.

DETAILED DESCRIPTION:
Allogeneic Transplantation and the Graft versus Disease Effect Over the past three decades, the transplantation of allogeneic marrow grafts has emerged as a uniquely effective therapy for patients with hematologic malignancies, marrow failure syndromes, and other lethal genetic and acquired diseases of hematopoiesis.1-9 Allogeneic transplantation potentially results in curative outcomes for patients with acute leukemia, chronic myelogenous leukemia, aplastic anemia, and lymphoid malignancies for whom standard therapies may not be effective. The anti-tumor effect mediated by allogeneic lymphocytes is an essential factor in eliminating residual disease post-transplant and preventing subsequent relapse.10-14 Numerous observations in patients undergoing allogeneic bone marrow transplant for hematological malignancies have convincingly demonstrated evidence of a graft-versus-disease (GVD) effect mediated by lymphocytes present in the donor graft. Supportive evidence for the importance of this phenomenon includes: 1) relapse rates of syngeneic BMT recipients are greater than in allogeneic recipients; 2) allogeneic BMT recipients who do not develop graft-versus-host disease (GVHD) have a significantly greater relapse rate than allogeneic BMT-recipients who do develop GVHD; 3) complete remissions have been observed in patients with relapsed disease after allogeneic BMT in association with flares of GVHD; 4) recipients of T-cell depleted BMT, a method of GVHD prophylaxis, relapse more frequently than recipients of non-T-cell depleted BMT; and 5) the use of an unrelated marrow graft in both non-T-cell depleted and T-cell depleted allogeneic BMT is associated with a reduced incidence of relapse.

The most direct evidence for the role of allogeneic lymphocytes in mediating an antitumor effect has been that patients who experience relapse following allogeneic transplantation may be successfully treated by the infusion of donor leukocytes.15-22 Summarizing the European experience, Kolb et al reported that the over 80% of patients with CML who relapse into the chronic phase following transplant may achieve a second complete remission after the infusion of donor leukocytes infusion in treating relapsed CML following transplant. Complete remissions with the use of DLI for the treatment of relapsed acute leukemias, chronic lymphocytic leukemia, myelodysplastic syndromes, multiple myeloma, and polycythemia vera, although lower than those seen in CML, have been well demonstrated by several groups. Additionally, a potent graft versus disease effect associated with allogeneic transplantation and donor leukocyte infusion has been observed in patients with non-Hodgkin's lymphoma and multiple myeloma.23-25 Thus, allogeneic transplantation offers a uniquely effective approach to eradicating hematological malignancy in which myeloablative therapy results in profound tumor cytoreduction and donor lymphocytes subsequently eliminate minimal residual disease via immunological mechanisms.

Limitations in the Application of Allogeneic Transplantation The use of allogeneic BMT has been limited by the significant treatment related morbidity and mortality associated with this procedure. Patients often experience significant organ dysfunction as a result of regimen related toxicity. Moderate to severe graft versus host disease occurs in approximately 40% of patients undergoing matched sibling conventional transplants and increases in incidence in older patients and those receiving unrelated or mismatched grafts.26-28 Opportunistic infections due to immune dysfunction remains a major source of morbidity and mortality particularly in older patients. The application of allogeneic transplantation is therefore restricted to younger patients with normal underlying organ function. Because the median age of many hematological malignancies may exceed 60 years of age, a majority of patients with these disorders are not considered candidates for this procedure.

The difficulty in applying allogeneic transplantation in patients with hematological malignancies is particularly highlighted in patients with lymphoid malignancies such as multiple myeloma, chronic lymphocytic leukemia and low-grade lymphoma. These disorders are incurable with standard dose chemotherapy but may follow a relatively indolent course for several years before patients develop progressive chemoresistant disease. Allogeneic transplantation has been associated with long-term disease free survival in these settings but is associated with a high incidence of upfront transplant related mortality. Strategies to limit transplant related toxicity are essential to translate the decreased incidence of relapse into an improvement in overall survival in this patient population.

Nonmyeloablative Allogeneic Transplantation One approach to limit the toxicity of allogeneic transplantation has been the use of nonmyeloablative regimens preceding the infusion of allogeneic cells.29-33 With this strategy, patients receive immunosuppressive therapy that allows for the engraftment of donor cells without the immediate eradication of patient hematopoiesis. The primary mechanism by which the underlying disease is eradicated is not through chemotherapy-mediated cytoreduction, but rather through the donor lymphocyte mediated graft versus tumor effect. As a result, patients experience far less regimen related toxicity. Therefore, the adoption of this strategy may allow for the use of allogeneic transplantation in disease settings and patient populations for which it had not been readily applicable in the past.

Over the past several years, the use nonmyeloablative transplant has rapidly expanded. Several reduced intensity conditioning regimens have been developed including fludarabine and cyclophosphamide; fludarabine and melphalan; fludarabine, anti-thymocyte globulin and low dose busulfan; and fludarabine and low dose TBI. Investigators have demonstrated the feasibility of this treatment approach with the majority of patients demonstrating donor engraftment, decreased regimen related toxicity, and graft mediated regression of disease. In some studies, patients demonstrate a period of mixed donor/host chimerism in which the infusion of donor lymphocytes is associated with achievement of complete donor chimerism.

Although regimen related toxicity is decreased following reduced intensive conditioning regimens, graft versus host disease and opportunistic infections remain a significant source of morbidity and mortality following nonmyeloablative allogeneic transplantation. The impact of nonmyeloablative transplantation on immunological reconstitution has not been fully defined. Persistence of host antigen presenting cells in the post-transplant period may increase the incidence of GVHD due to the presentation of alloantigens to donor T cells. In contrast, residual host cellular immunity may provide enhanced protection against infectious pathogens and allow for more rapid education of donor lymphocytes. Of note, CMV infections remain common in this population but present later in the post-transplant period characteristically following the attainment of full donor chimerism.34

Nonmyeloablative Allogeneic Transplantation in Conjunction with CAMPATH Therapy One approach to reduce the incidence of GVHD following nonmyeloablative transplantation is the addition of CAMPATH to the preparative regimen to deplete T cells from both the recipient and the incoming graft.35 CAMPATH-1H (Alemtuzumab) is a recombinant DNA-derived humanized monoclonal antibody directed against the cell surface glycoprotein, CD52; produced in mammalian cell (Chinese hamster ovary) suspension.36-39 Campath-1H is indicated for the treatment of B-cell chronic lymphocytic leukemia in patients who have been treated with alkylating agents and have failed fludarabine therapy. Campath-1H has been used in patients with autoimmune neutropenia, non-Hodgkin's lymphoma, rheumatoid arthritis, and vasculitis. It has also been used to prevent graft-versus-host disease in patients receiving stem cell transplantation. GVHD prophylaxis was with cyclosporin A alone.

Mackinnon et al investigated a nonmyeloablative conditioning regimen in 47 patients with hematological malignancies receiving allogeneic bone marrow stem cells from matched, unrelated donors.40 The majority of patients had high-risk features, including having failed a prior transplantation (29 individuals). Twenty of the transplants were mismatched for HLA class I and/or class II alleles. They added CAMPATH-1H to a preparative regimen of fludarabine and melphalan and administered either GCSF mobilized peripheral blood stems or unmanipulated bone marrow from matched unrelated donors. Primary graft failure occurred in only 2 of 44 evaluable patients (4.5%). Chimerism studies in 34 patients indicated that the majority (85.3%) attained initial full donor chimerism. Only 3 patients developed grade III to IV acute GVHD, and no patients have yet developed chronic extensive GVHD. The estimated probability of nonrelapse mortality at day 100 was 14.9% (95% confidence interval [CI], 4.7%-25.1%). With a median follow-up of 344 days (range, 79-830), overall and progression-free survivals at 1 year were 75.5% (95% CI, 62.8%-88.2%) and 61.5% (95% CI, 46.1%-76.8%), respectively. It was subsequently reported that a significant subset of patients demonstrated evidence of CMV reactivation.41 However, the presence of CMV did not negatively impact survival. While the investigators noted a need for longer follow-up of this cohort, they felt that this preparative regimen incorporating in vivo CAMPATH-1H was associated with durable engraftment and minimal treatment related toxicity.

Immune Reconstitution Following Allogeneic Transplantation Allogeneic transplantation is associated with a period of immune dysfunction that characteristically persists for at least 1 year post-transplant.42,43 Immune recovery is dependent on the reconstitution of elements of humoral and cellular immunity and their reeducation in the transplant recipient. It is particularly delayed in recipients of an unrelated or T cell depleted graft. The post-transplant period is characterized by decreased levels of helper T cells, an associated inversion of the C4:CD8 ratio, and the blunting of T cell responses to mitogenic stimuli and recall antigens.44-46 Humoral immune dysfunction is associated with the loss of protective antibody levels to bacterial and viral pathogens, decreased levels of circulating immunoglobulins particularly of the IgG2 subtype, and the reduced complexity in the pattern of the immunoglobulin gene rearrangement.47,48

Dendritic Cells and Immune Reconstitution The nature of the recovery of antigen presenting cells such as dendritic cells are likely to play an essential role in the reconstitution of posttransplant immunity and host/donor tolerance. Dendritic cells (DC) form a complex network of antigen presenting cells that play a vital role in the induction of primary immunity as well as the modulation of tolerance.49.50 DC are the most potent antigen presenting cells and are uniquely able to induce primary immune responses against novel antigens through the rich expression of costimulatory and adhesion molecules. DC generated from nonmyeloid lineages or in an immature state may mediate immune tolerance and direct T cell responses towards a TH2 phenotype. Distinct DC populations have been identified in the peripheral blood that are differentiated by the presence of myeloid (CD11c) or plasmacytoid (CD123) markers.51,52 DC2 (plasmacytoid) cells are characterized by expression of type 2 cytokines and thus initiate a Th2 response, whereas DC1 (myeloid) cells initiate Th1 cytokine response. DC isolated from patients with malignancy demonstrate functional deficiencies that potentially contribute to lack of tumor recognition by host immunity. Little is known about DC engraftment or phenotypic and functional characteristics after allogeneic transplantation. The interactions of DC with effector populations is likely to be unique following nonmyeloablative conditioning given the presence of mixed donor/recipient chimerism that may characterize the post-transplant period.

In a murine model, Shlomchik et al demonstrated that persistence of host antigen presenting cells post-transplant was associated with the development of GVHD.53 In this model, host DC capable of presenting minor histocompatibility antigens to infused donor T-cells potentially initiate T-cell activation and an associated Th-1 cytokine cascade implicated in the pathogenesis of aGVHD. The relative levels of DC1/DC2 subsets in the hematopoietic graft strongly correlate with the incidence of graft versus host disease and incidence of relapse. G-CSF mediated stem mobilization is associated with increased levels of DC2 populations.54 In an animal model, the infusion of splenocytes and bone marrow from donors treated with G-CSF was associated with emergence of a DC2 phenotype, and thus, tolerance.55 In one study of patients undergoing allogeneic transplantation, the presence of increased numbers of DC2 cells in the hematopoietic graft was associated with a decrease in GVHD, and increase in relapse and poorer outcomes.56 The impact of DC chimerism, patterns of reconstitution, and presence of DC1 and DC2 populations following nonmyeloablative allogeneic transplantation has not been well studied. Recent studies have demonstrated that CD52 is expressed by some DC populations and suggest that CAMPATH therapy may impact antigen presentation by depletion of DC populations from the host.57-59 Depletion of host derived DC may decrease in the incidence of GVHD, while presence of donor DC is likely essential for the reconstitution of cellular immunity.

In the proposed study, we intend to examine the application of a CAMPATH based preparative regimen in patients with hematological malignancies undergoing nonmyeloablative allogeneic stem cell transplantation from an unrelated donor. The study will involve patients who would otherwise not be candidates for a conventional myeloablative conditioning regimen because of age or organ dysfunction and who do not have HLA-matched sibling donors. It will also include patients suffering from lymphoid malignancies such as low-grade lymphoma, CLL, and multiple myeloma that have experienced unacceptably high transplant related mortality with conventional allogeneic transplantation. Inclusion of both myeloid and lymphoid hematological malignancies in the study cohort will optimize accrual and will not limit the ability to the ability to pursue the study goals. Patterns of engraftment, graft versus host disease, immune reconstitution, and donor/host chimerism are primarily determined by the preparative regimen and transplant strategy and should not differ considerably within the patient cohort.

For the conditioning regimen, we have chosen an intermediate dose of cyclophosphamide and fludarabine in an attempt to minimize the incidence of graft rejection without increasing the frequency of treatment related morbidity and mortality. Based on the work of MacKinnon et al, we will add CAMPATH-1H to the preparative regimen to further decrease the incidence of GVHD and promote donor stem cell engraftment. Following this regimen circulating levels CAMPATH are present for several weeks post-transplant and may excessively deplete donor T cells as well as eliminate DC populations from the donor graft. In an effort to improve post-transplant immune reconstitution and limit risks of infection and relapse, we have chosen a lower dose of CAMPATH and will follow levels at serial time points post-transplant.

The principal endpoints of the trial will include defining: 1) the treatment related toxicity profile and post-transplant hematopoietic recovery 2) the incidence and severity of CMV infection and acute and chronic GVHD 3) the phenotypic and functional characteristics of DC and T cell populations post-transplant; and 4) the patterns of donor/host chimerism in DC and T cell populations and its correlation with GVHD. As a secondary endpoint, 1 and 2 year DFS and OS will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 65 years. There is no lower age limit. Patients 65 years and older will be accrued on a case-by-case basis to this protocol, after discussion and approval by the principal investigator. The acceptance to this protocol for such patients would be based on the absence of coexisting medical problems, which would seriously compromise the patient's ability to tolerate the known morbidity and risks of bone marrow transplantation.
* Patients must have a 5/6 or 6/6 HLA matched, unrelated donor of bone marrow stem cells.
* Each patient must be willing to participate as a research subject and must sign an informed consent form after having been advised as to the nature and risk of the study prior to entering the protocol. Parents or legal guardians of patients who are minors will sign the informed consent form after being advised of the nature and risks of the study. Attending physicians in the Bone Marrow Transplant Service will enroll patients to this study and will obtain written consents.

Eligibility Criteria - Donor

* 5/6 or 6/6 HLA matched with the recipient as determined by molecular testing. Donors will be identified through the National Marrow Donor Program for unrelated donors.
* Donor selection will be performed as outlined in the donor selection SOP's. In patients who have more than one potential donor preference will be given to donors who have no evidence of CMV exposure (if the recipient is CMV-), those who are younger and those who are male. Selection of an unrelated donor from the NMDP registry will proceed according to the donor selection SOP. Molecular testing of HLA-A, B, and DR alleles will identify potential donors and the American Red Cross HLA lab will confirm all typing. Donor selection will be coordinated with transplant physician and the HLA laboratory director. Preference will be given to donors who are 6/6 molecular matches, those who are CMV- (if the recipient is CMV-), those who are younger, and males.

Exclusion Criteria:

* Active CNS leukemia involvement.
* Female patients who are pregnant or breast feeding
* Karnofsky performance status < 70%, (appendix 1).
* Left ventricular ejection fraction of < 40%.
* Serum creatinine > 1.5 X normal
* Patients seropositive for HIV; HTLV -1, or with evidence of chronic active hepatitis as demonstrated by detection of hepatitis surface antigen in the serum
* Patients with serologic evidence of hepatitis B or C exposure will undergo liver biopsy to assess for presence of active hepatitis or fibrosis and quantification of risk of proceeding with transplant
* Patients not providing informed consent.
* Patients with known hypersensitivity to E. Coli derived products.
* SGOT and SGPT > 2.5 x ULN, unless thought to be disease related
* Total bilirubin > 2.0 mg/dl, with direct bilirubin > 0.5 mg/dl

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2002-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Primary objective of study is to determine the safety of non-myeloablative allogenic stem cell transplantation from matched unrelated donors in patients with hematologic malignancies with a focus on the incidence of treatment-related mortality. | Within 100 days of transplant

SECONDARY OUTCOMES:
Secondary clinical endpoints includes; incidence of graft failure or rejection; incidence and severity of acute and chronic GVHD; tumor response, and long-term overall and disease-free survival. | Within 100 days of transplant

CONTACTS AND LOCATIONS:
Overall Officials: David F McDermott, MD, Principal Investigator — Beth Israel Deaconess Medical Center; David E Avigan, MD, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States